CLINICAL TRIAL: NCT05603403
Title: Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Trial Placebo-Controlled Clinical Trial To Evaluate The Efficacy And Safety Of Probiatop In The Treatment Of Digestive Symptoms
Brief Title: Efficacy And Safety Of Probiatop In The Treatment Of Digestive Symptoms
Acronym: Probiatop
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Collaborators: Farmoquimica S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROFQM0422OR-IV; 60215522.6.1001.5412 (Other: CAAE)
Record Dates: First submitted 2022-10-20; First posted 2022-11-02 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Signs and Symptoms, Digestive
Keywords: Signs and Symptoms Digestive; Probiatop; Digestive Symptoms
MeSH Terms: conditions — Signs and Symptoms, Digestive | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Investigational product (Probiatop) and Placebo
Who Masked: Participant, Investigator
Masking Description: The study will be double-blind. The participants and the investigator will be "blinded" in the study, in which they will not know the treatment that each participant will be receiving.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiatop (Experimental): Probiotic used in the reconstitution and rebalancing of the intestinal microbiota.
  Association of probiotic strains containing 1 g/sachet of 1 x 109 Bifidobacterium lactis HN019, 1 x 109 Lactobacillus acidophilus, 1 x 109 Lactobacillus rhamnosus HN001 / Lacticaseibacillus rhamnosus HN001 and 1 x 109 Lactobacillus paracasei Lpc- 37 / Lacticaseibacillus paracasei Lpc-37.
  Interventions: Drug: Probiatop
- Hydrolized collagen (Placebo Comparator): Hydrolyzed collagen is approved by Agência Nacional de Vigilância Sanitária (ANVISA) including for use in infants (ANVISA, IN NO. 28, OF JULY 26, 2018). Its use as a placebo is convenient, as it dissolves well in water, and promotes good masking. Based on literature surveys on hydrolyzed collagen and the intestinal microbiota, it was verified that the dose used (1 g) would not promote relevant functional impact in the context of the habitual Brazilian people diet.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Probiatop — 1 sachet orally, 2 times a day, for 42 days
  Other Names: Probiotic
  Arms: Probiatop
Other: Placebo — 1 sachet orally, 2 times a day, for 42 days
  Other Names: Placebo Comparator
  Arms: Hydrolized collagen

SUMMARY:
A Multicenter, Randomized, Double-blind, Placebo-Controlled Clinical Trial to Evaluate the Efficacy and Safety of Probiatop in the Treatment of Digestive Symptoms. Phase IV. The casuistic presented in this protocol is 150 participants randomized at a 1:1 ratio (75 receiving Probiatop and 75 receiving placebo), balanced by age, sex, prebiotic intake* and summation of the Gastrointestinal Symptom Rating Scale (GSRS) questions related to the domains of diarrhea (questions 11, 12, and 14), indigestion (questions 6, 7, 8, and 9), and constipation (questions 10, 13, and 15) separated by intensity and frequency. Participants with recurrent digestive symptoms for at least 3 months, with a score of 21 on the sum of questions 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15 of the GSRS (corresponding to the domains diarrhea, indigestion and constipation) will be randomized to Probiatop or placebo.

DETAILED DESCRIPTION:
This is a Phase IV clinical trial that will evaluate the efficacy and safety of Probiatop (investigational product). Participants with recurrent digestive symptoms for at least 3 months, with a score of 21 on the sum of questions: 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15 of the GSRS questionnaire (corresponding to the domains diarrhea, indigestion and constipation) will be randomized to Probiatop or placebo. It will also be applied by electronic means (whatsapp link) on D7, D21 and D35. On these days participants will also be contacted by telemedicine to collect adverse events adverse events and data on concomitant medication. Treatment will be discontinued on D42. On D70 the participant will again be contacted by telemedicine for final data collection.

Product under investigation and dosage: Probiatop composition: association of probiotic strains containing 1 g/sachet of 1 x 109 CFU Bifidobacterium lactis HN019 (ATCC SD 5674), 1 x 109 CFU Lactobacillus acidophilus NCFM (ATCC SD 5221), 1 x 109 CFU Lactobacillus rhamnosus HN001 / Lacticaseibacillus rhamnosus HN001 (ATCC SD 5675) and 1 x 109 CFU Lactobacillus paracasei Lpc-37 / Lacticaseibacillus paracasei Lpc-37 (ATCC SD 5275). Placebo composition: collagen

ELIGIBILITY:
Inclusion Criteria:

* Male or female gender;
* Age ≥ 18 years;
* BMI ≥ 18, 5 ≤ 29.9 Kg/m2;
* Complaint of recurrent digestive symptoms for at least 3 months with value ≥ 21 of the sum of questions: 6, 7, 8, 9, 10, 11, 12, 13, 14, and 15 of the GSRS in frequency or intensity separately.

Exclusion Criteria:

* Extreme eating habits for which the primary intervention is dietary re-education: more than 7 of the of the 14 main meals of the week (lunch and dinner) based on ultra-processed products (industrial formulations formulations such as: filled cookies, "packaged" snacks packaged" snacks, soft drinks and "instant" noodles, frozen frozen and ready-to-eat products such as pasta, pizzas hamburgers, nuggets, sausages, etc) or "fast food" or average consumption of soft drinks exceeding 2 glasses per day.
* Alcoholism (DSM V): disorder defined as the repetition problems resulting from the use of alcohol that lead to clinically significant clinically significant impairment and/or suffering;
* Diabetes mellitus type I or II;
* Chronic diarrhea with signs of malabsorption (weight loss bulky and exceptionally smelly stools), AND/OR bleeding, AND/OR presence of mucus in the stool, bleeding without diarrhea;
* Weight loss ≥ 10% in the past 6 months;
* Any recent change in eating habit, including veganism;
* Clinically significant illnesses at the discretion of the Investigator;
* Use of medications or supplements that may modify gastrointestinal function in the 30 days prior to randomization, especially proton pump inhibitors antacids, laxatives, constipating agents (loperamide, racecadotrilla, tricyclic antidepressants), other probiotics and prebiotics (containing dietary fiber including inulin, resistant starch, cellulose, oligofructose, fiber oligofructose, soy fiber, polydextrose, Kefir, Kombucha, and others);
* Use of antibiotics in the 3 months prior to randomization for any indications, including Helicobacter pylori;
* History of digestive surgery;
* Active cancer or cancer under treatment in the 6 months prior to randomization, except operated basal cell carcinoma;
* History of allergy or hypersensitivity to probiotics or components of the formula;
* Pregnant and lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Clinical Outcome Measure: Efficacy | 42 days
  Multicriteria evaluation of the impact of Probiatop on gastrointestinal symptom reduction symptoms by the Gastrointestinal Symptom Rating Scale (GSRS).

SECONDARY OUTCOMES:
Clinical Outcome Measure: Safety | 42 days
  Evaluation of the impact of Probiatop on the reduction of each domain of the questionnaire Gastrointestinal Symptom Rating Scale (GSRS) - abdominal pain, reflux syndrome, diarrhea, indigestion and constipation.
Clinical Outcome Measure: Safety | Day 0 to Day 42
  Incidence and severity of adverse reactions to Probiatop.

CONTACTS AND LOCATIONS:
Overall Officials: Regina Mayumi Doi, MD, Principal Investigator — A2Z CLINICAL CENTRO AVANCADO DE PESQUISA CLINICA EIRELI
Locations (1):
- A2Z Clinical Centro Avancado de Pesquisa Clinica Eireli, Valinhos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
It is believed that after the data analysis and presentation to the National Commission on Research Ethics, all data will become public.

REFERENCES:
- [Background] ANVISA, Instrução Normativa - IN Nº 28, DE 26 DE JULHO DE 2018. Estabelece as listas de constituintes, de limites de uso, de alegações e de rotulagem complementar dos suplementos alimentares. Almeida, L. B., C. B. Marinho, C. S. Souza and V. Cheib (2009).
- [Background] Almeida, L. B., C. B. Marinho, C. S. Souza and V. Cheib (2009).
- [Background] Bae JY, Kim JI, Park S, Yoo K, Kim IH, Joo W, Ryu BH, Park MS, Lee I, Park MS. Effects of Lactobacillus plantarum and Leuconostoc mesenteroides Probiotics on Human Seasonal and Avian Influenza Viruses. J Microbiol Biotechnol. 2018 Jun 28;28(6):893-901. doi: 10.4014/jmb.1804.04001. PMID 29847863
- [Background] Blumstein DT, Levy K, Mayer E, Harte J. Gastrointestinal dysbiosis. Evol Med Public Health. 2014;2014(1):163. doi: 10.1093/emph/eou029. Epub 2014 Nov 20. No abstract available. PMID 25416734
- [Background] Breton J, Galmiche M, Dechelotte P. Dysbiotic Gut Bacteria in Obesity: An Overview of the Metabolic Mechanisms and Therapeutic Perspectives of Next-Generation Probiotics. Microorganisms. 2022 Feb 16;10(2):452. doi: 10.3390/microorganisms10020452. PMID 35208906
- [Background] Chen Y, Zhou J, Wang L. Role and Mechanism of Gut Microbiota in Human Disease. Front Cell Infect Microbiol. 2021 Mar 17;11:625913. doi: 10.3389/fcimb.2021.625913. eCollection 2021. PMID 33816335
- [Background] Cremonini F, Di Caro S, Nista EC, Bartolozzi F, Capelli G, Gasbarrini G, Gasbarrini A. Meta-analysis: the effect of probiotic administration on antibiotic-associated diarrhoea. Aliment Pharmacol Ther. 2002 Aug;16(8):1461-7. doi: 10.1046/j.1365-2036.2002.01318.x. PMID 12182746
- [Background] Cruchet S, Furnes R, Maruy A, Hebel E, Palacios J, Medina F, Ramirez N, Orsi M, Rondon L, Sdepanian V, Xochihua L, Ybarra M, Zablah RA. The use of probiotics in pediatric gastroenterology: a review of the literature and recommendations by Latin-American experts. Paediatr Drugs. 2015 Jun;17(3):199-216. doi: 10.1007/s40272-015-0124-6. PMID 25799959
- [Background] de Almada CN, Nunes de Almada C, Martinez RC, Sant'Ana Ade S. Characterization of the intestinal microbiota and its interaction with probiotics and health impacts. Appl Microbiol Biotechnol. 2015 May;99(10):4175-99. doi: 10.1007/s00253-015-6582-5. Epub 2015 Apr 21. PMID 25895093
- [Background] Ding RX, Goh WR, Wu RN, Yue XQ, Luo X, Khine WWT, Wu JR, Lee YK. Revisit gut microbiota and its impact on human health and disease. J Food Drug Anal. 2019 Jul;27(3):623-631. doi: 10.1016/j.jfda.2018.12.012. Epub 2019 Feb 1. PMID 31324279
- [Background] Divella R, DE Palma G, Tufaro A, Pelagio G, Gadaleta-Caldarola G, Bringiotti R, Paradiso A. Diet, Probiotics and Physical Activity: The Right Allies for a Healthy Microbiota. Anticancer Res. 2021 Jun;41(6):2759-2772. doi: 10.21873/anticanres.15057. PMID 34083266
- [Background] Fan Y, Pedersen O. Gut microbiota in human metabolic health and disease. Nat Rev Microbiol. 2021 Jan;19(1):55-71. doi: 10.1038/s41579-020-0433-9. Epub 2020 Sep 4. PMID 32887946
- [Background] Ford AC, Harris LA, Lacy BE, Quigley EMM, Moayyedi P. Systematic review with meta-analysis: the efficacy of prebiotics, probiotics, synbiotics and antibiotics in irritable bowel syndrome. Aliment Pharmacol Ther. 2018 Nov;48(10):1044-1060. doi: 10.1111/apt.15001. Epub 2018 Oct 8. PMID 30294792
- [Background] Fraher MH, O'Toole PW, Quigley EM. Techniques used to characterize the gut microbiota: a guide for the clinician. Nat Rev Gastroenterol Hepatol. 2012 Mar 27;9(6):312-22. doi: 10.1038/nrgastro.2012.44. PMID 22450307
- [Background] Ganji-Arjenaki M, Rafieian-Kopaei M. Probiotics are a good choice in remission of inflammatory bowel diseases: A meta analysis and systematic review. J Cell Physiol. 2018 Mar;233(3):2091-2103. doi: 10.1002/jcp.25911. Epub 2017 May 3. PMID 28294322
- [Background] Gebrayel P, Nicco C, Al Khodor S, Bilinski J, Caselli E, Comelli EM, Egert M, Giaroni C, Karpinski TM, Loniewski I, Mulak A, Reygner J, Samczuk P, Serino M, Sikora M, Terranegra A, Ufnal M, Villeger R, Pichon C, Konturek P, Edeas M. Microbiota medicine: towards clinical revolution. J Transl Med. 2022 Mar 7;20(1):111. doi: 10.1186/s12967-022-03296-9. PMID 35255932
- [Background] Hill C, Guarner F, Reid G, Gibson GR, Merenstein DJ, Pot B, Morelli L, Canani RB, Flint HJ, Salminen S, Calder PC, Sanders ME. Expert consensus document. The International Scientific Association for Probiotics and Prebiotics consensus statement on the scope and appropriate use of the term probiotic. Nat Rev Gastroenterol Hepatol. 2014 Aug;11(8):506-14. doi: 10.1038/nrgastro.2014.66. Epub 2014 Jun 10. PMID 24912386
- [Background] Houghteling PD, Walker WA. Why is initial bacterial colonization of the intestine important to infants' and children's health? J Pediatr Gastroenterol Nutr. 2015 Mar;60(3):294-307. doi: 10.1097/MPG.0000000000000597. PMID 25313849
- [Background] Huang R, Wang K, Hu J. Effect of Probiotics on Depression: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Nutrients. 2016 Aug 6;8(8):483. doi: 10.3390/nu8080483. PMID 27509521
- [Background] Johnston BC, Lytvyn L, Lo CK, Allen SJ, Wang D, Szajewska H, Miller M, Ehrhardt S, Sampalis J, Duman DG, Pozzoni P, Colli A, Lonnermark E, Selinger CP, Wong S, Plummer S, Hickson M, Pancheva R, Hirsch S, Klarin B, Goldenberg JZ, Wang L, Mbuagbaw L, Foster G, Maw A, Sadeghirad B, Thabane L, Mertz D. Microbial Preparations (Probiotics) for the Prevention of Clostridium difficile Infection in Adults and Children: An Individual Patient Data Meta-analysis of 6,851 Participants. Infect Control Hosp Epidemiol. 2018 Jul;39(7):771-781. doi: 10.1017/ice.2018.84. Epub 2018 Apr 26. PMID 29695312
- [Background] Khurshid M, Aslam B, Nisar MA, Akbar R, Rahman H, Khan AA, Rasool MH. Bacterial munch for infants: potential pediatric therapeutic interventions of probiotics. Future Microbiol. 2015;10(11):1881-95. doi: 10.2217/fmb.15.102. Epub 2015 Oct 30. PMID 26515509
- [Background] Kopp-Hoolihan L. Prophylactic and therapeutic uses of probiotics: a review. J Am Diet Assoc. 2001 Feb;101(2):229-38; quiz 239-41. doi: 10.1016/S0002-8223(01)00060-8. PMID 11271697
- [Background] Kurugol Z, Koturoglu G. Effects of Saccharomyces boulardii in children with acute diarrhoea. Acta Paediatr. 2005 Jan;94(1):44-7. doi: 10.1111/j.1651-2227.2005.tb01786.x. PMID 15858959
- [Background] Lange K, Buerger M, Stallmach A, Bruns T. Effects of Antibiotics on Gut Microbiota. Dig Dis. 2016;34(3):260-8. doi: 10.1159/000443360. Epub 2016 Mar 30. PMID 27028893
- [Background] Li D, Wang P, Wang P, Hu X, Chen F. The gut microbiota: A treasure for human health. Biotechnol Adv. 2016 Nov 15;34(7):1210-1224. doi: 10.1016/j.biotechadv.2016.08.003. Epub 2016 Aug 31. PMID 27592384
- [Background] Linares DM, Ross P, Stanton C. Beneficial Microbes: The pharmacy in the gut. Bioengineered. 2016;7(1):11-20. doi: 10.1080/21655979.2015.1126015. PMID 26709457
- [Background] Marchesi JR, Adams DH, Fava F, Hermes GD, Hirschfield GM, Hold G, Quraishi MN, Kinross J, Smidt H, Tuohy KM, Thomas LV, Zoetendal EG, Hart A. The gut microbiota and host health: a new clinical frontier. Gut. 2016 Feb;65(2):330-9. doi: 10.1136/gutjnl-2015-309990. Epub 2015 Sep 2. PMID 26338727
- [Background] Revicki DA, Wood M, Wiklund I, Crawley J. Reliability and validity of the Gastrointestinal Symptom Rating Scale in patients with gastroesophageal reflux disease. Qual Life Res. 1998 Jan;7(1):75-83. doi: 10.1023/a:1008841022998. PMID 9481153
- [Background] Sanchez B, Delgado S, Blanco-Miguez A, Lourenco A, Gueimonde M, Margolles A. Probiotics, gut microbiota, and their influence on host health and disease. Mol Nutr Food Res. 2017 Jan;61(1). doi: 10.1002/mnfr.201600240. Epub 2016 Oct 10. PMID 27500859
- [Background] Sanders ME, Heimbach JT, Pot B, Tancredi DJ, Lenoir-Wijnkoop I, Lahteenmaki-Uutela A, Gueimonde M, Banares S. Health claims substantiation for probiotic and prebiotic products. Gut Microbes. 2011 May-Jun;2(3):127-33. doi: 10.4161/gmic.2.3.16174. Epub 2011 May 1. PMID 21646865
- [Background] Souza GS, Sarda FA, Giuntini EB, Gumbrevicius I, Morais MB, Menezes EW. TRANSLATION AND VALIDATION OF THE BRAZILIAN PORTUGUESE VERSION OF THE GASTROINTESTINAL SYMPTOM RATING SCALE (GSRS) QUESTIONNAIRE. Arq Gastroenterol. 2016 Jul-Sep;53(3):146-51. doi: 10.1590/S0004-28032016000300005. PMID 27438418
- [Background] Thaiss CA, Itav S, Rothschild D, Meijer MT, Levy M, Moresi C, Dohnalova L, Braverman S, Rozin S, Malitsky S, Dori-Bachash M, Kuperman Y, Biton I, Gertler A, Harmelin A, Shapiro H, Halpern Z, Aharoni A, Segal E, Elinav E. Persistent microbiome alterations modulate the rate of post-dieting weight regain. Nature. 2016 Dec 22;540(7634):544-551. doi: 10.1038/nature20796. Epub 2016 Nov 24. PMID 27906159
- [Background] Turnbaugh PJ, Ley RE, Mahowald MA, Magrini V, Mardis ER, Gordon JI. An obesity-associated gut microbiome with increased capacity for energy harvest. Nature. 2006 Dec 21;444(7122):1027-31. doi: 10.1038/nature05414. PMID 17183312
- [Background] Turnbaugh PJ, Ridaura VK, Faith JJ, Rey FE, Knight R, Gordon JI. The effect of diet on the human gut microbiome: a metagenomic analysis in humanized gnotobiotic mice. Sci Transl Med. 2009 Nov 11;1(6):6ra14. doi: 10.1126/scitranslmed.3000322. PMID 20368178
- [Background] Vandenplas Y, Huys G, Daube G. Probiotics: an update. J Pediatr (Rio J). 2015 Jan-Feb;91(1):6-21. doi: 10.1016/j.jped.2014.08.005. Epub 2014 Oct 23. PMID 25458874
- [Background] Waskito LA, Rezkitha YAA, Vilaichone RK, Wibawa IDN, Mustika S, Sugihartono T, Miftahussurur M. Antimicrobial Resistance Profile by Metagenomic and Metatranscriptomic Approach in Clinical Practice: Opportunity and Challenge. Antibiotics (Basel). 2022 May 13;11(5):654. doi: 10.3390/antibiotics11050654. PMID 35625299
- [Background] Wei L, Singh R, Ro S, Ghoshal UC. Gut microbiota dysbiosis in functional gastrointestinal disorders: Underpinning the symptoms and pathophysiology. JGH Open. 2021 Mar 23;5(9):976-987. doi: 10.1002/jgh3.12528. eCollection 2021 Sep. PMID 34584964